CLINICAL TRIAL: NCT01067703
Title: Remote Ischaemic Preconditioning for Heart Surgery
Brief Title: Remote Ischaemic Preconditioning for Heart Surgery (RIPHeart-Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: German Research Foundation (Other); Goethe University (Other)
Responsible Party: Principal Investigator, Patrick Meybohm, Prof. Dr. Patrick Meybohm, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ME 3559/1-1
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Injury; Mortality
Keywords: remote ischaemic preconditioning, cardiac surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC (Active Comparator)
  Interventions: Procedure: Remote Ischemic Preconditioning
- CONTROL (Sham Comparator)
  Interventions: Procedure: Control/sham procedure (blood pressure cuff)

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — RIPC will be induced during anesthesia by four 5-min cycles of upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200 mm Hg, whereas the pressure has to be at least 20 mm Hg greater than the systolic arterial pressure measured via the arterial line.
  Arms: RIPC
Procedure: Control/sham procedure (blood pressure cuff) — Sham placement of the blood pressure cuff around a dummy arm inflated to a pressure of 200 mm Hg with four cycles of 5 min inflation and 5 min deflation.
  Arms: CONTROL

SUMMARY:
The purpose of this study is to evaluate the effects of Remote Ischaemic Preconditioning on perioperative ischaemic injury in patients undergoing cardiac surgery compared to control intervention.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass is associated with a predictable incidence of myocardial, neurological and renal dysfunction. This significant morbidity and mortality is at least partly due to perioperative ischaemia. Remote ischaemic preconditioning (RIPC) is a novel, simple, non-invasive and inexpensive intervention by which ischaemia of non-vital tissue (skeletal muscles) protects remote organs (heart, brain and kidney) from a subsequent sustained episode of ischaemia. The investigators perform a multicenter randomized controlled study to evaluate that RIPC reduces teh severity of perioperative ischaemic injury in patients undergoing cardiac surgery, and results in about 1/3 risk reduction in the occurence of major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing heart surgery on cardiopulmonary bypass

Exclusion Criteria:

* age < 18
* Emergency cases
* left ventricular ejection fraction less than 30%
* current atrial fibrillation
* Inability to give informed consent
* preoperative use of inotropics or mechanical assist device
* severe liver, renal and pulmonary disease
* recent myocardial infarction (within 7 days)
* recent systemic infection or sepsis (within 7 days)
* severe stroke (within 2 months)
* peripheral vascular disease affecting upper limbs
* previous serious psychiatric disorders (e.g. schizophrenia, dementia)
* concomitant carotid endarterectomy
* rare surgeries: cardiac transplantation, correction of complicated congenital anomalies, pulmonary thromboembolectomy, off-pump surgery, minimal-invasive operation without sternotomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, non-fatal myocardial infarction, any new stroke, and/or acute renal failure | In-hospital
  Time frame until hospital discharge

SECONDARY OUTCOMES:
Occurence of any component of the composite outcome | Postoperative hospital discharge, 3 months, 12 months
length of stay on the intensive care unit | Postoperative during hospital stay
total hospital stay | hospital discharge
new onset of atrial fibrillation | In-hospital
Delirium | Postoperative 24, 48, 72, 96 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, MD, Principal Investigator — University Hospital Frankfurt/ University Hospital Schleswig-Holstein; Berthold Bein, MD, DESA, Principal Investigator — University Hospital Schleswig-Holstein; Jochen Cremer, MD, Principal Investigator — University Hospital Schleswig-Holstein; Kai Zacharowski, MD, PhD, Principal Investigator — University Hospital Frankfurt am Main
Locations (10):
- Germany (10):
  - University Hospital Aachen (RWTH), Aachen
  - University Hospital Charite, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Frankfurt/M, Frankfurt/M
  - University Hospital Goettingen, Göttingen
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital of Schleswig-Holstein, Lübeck
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Rostock, Rostock
  - University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Result] Meybohm P, Bein B, Brosteanu O, Cremer J, Gruenewald M, Stoppe C, Coburn M, Schaelte G, Boning A, Niemann B, Roesner J, Kletzin F, Strouhal U, Reyher C, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Stehr SN, Kortgen A, Wittmann M, Baumgarten G, Meyer-Treschan T, Kienbaum P, Heringlake M, Schon J, Sander M, Treskatsch S, Smul T, Wolwender E, Schilling T, Fuernau G, Hasenclever D, Zacharowski K; RIPHeart Study Collaborators. A Multicenter Trial of Remote Ischemic Preconditioning for Heart Surgery. N Engl J Med. 2015 Oct 8;373(15):1397-407. doi: 10.1056/NEJMoa1413579. Epub 2015 Oct 5. PMID 26436208
- [Result] Meybohm P, Zacharowski K, Cremer J, Roesner J, Kletzin F, Schaelte G, Felzen M, Strouhal U, Reyher C, Heringlake M, Schon J, Brandes I, Bauer M, Knuefermann P, Wittmann M, Hachenberg T, Schilling T, Smul T, Maisch S, Sander M, Moormann T, Boening A, Weigand MA, Laufenberg R, Werner C, Winterhalter M, Treschan T, Stehr SN, Reinhart K, Hasenclever D, Brosteanu O, Bein B; RIP Heart-Study Investigator Group. Remote ischaemic preconditioning for heart surgery. The study design for a multi-center randomized double-blinded controlled clinical trial--the RIPHeart-Study. Eur Heart J. 2012 Jun;33(12):1423-6. PMID 22880214
- [Derived] Westphal S, Stoppe C, Gruenewald M, Bein B, Renner J, Cremer J, Coburn M, Schaelte G, Boening A, Niemann B, Kletzin F, Roesner J, Strouhal U, Reyher C, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Kortgen A, Stehr SN, Wittmann M, Baumgarten G, Struck R, Meyer-Treschan T, Kienbaum P, Heringlake M, Schoen J, Sander M, Treskatsch S, Smul T, Wolwender E, Schilling T, Degenhardt F, Franke A, Mucha S, Tittmann L, Kohlhaas M, Fuernau G, Brosteanu O, Hasenclever D, Zacharowski K, Meybohm P; RIPHeart-Study Collaborators. Genome-wide association study of myocardial infarction, atrial fibrillation, acute stroke, acute kidney injury and delirium after cardiac surgery - a sub-analysis of the RIPHeart-Study. BMC Cardiovasc Disord. 2019 Jan 24;19(1):26. doi: 10.1186/s12872-019-1002-x. PMID 30678657
- [Derived] Meybohm P, Kohlhaas M, Stoppe C, Gruenewald M, Renner J, Bein B, Albrecht M, Cremer J, Coburn M, Schaelte G, Boening A, Niemann B, Sander M, Roesner J, Kletzin F, Mutlak H, Westphal S, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Stehr SN, Kortgen A, Wittmann M, Baumgarten G, Meyer-Treschan T, Kienbaum P, Heringlake M, Schoen J, Treskatsch S, Smul T, Wolwender E, Schilling T, Fuernau G, Bogatsch H, Brosteanu O, Hasenclever D, Zacharowski K; RIPHeart (Remote Ischemic Preconditioning for Heart Surgery) Study Collaborators. RIPHeart (Remote Ischemic Preconditioning for Heart Surgery) Study: Myocardial Dysfunction, Postoperative Neurocognitive Dysfunction, and 1 Year Follow-Up. J Am Heart Assoc. 2018 Mar 26;7(7):e008077. doi: 10.1161/JAHA.117.008077. PMID 29581218
- [Derived] Candilio L, Malik A, Ariti C, Barnard M, Di Salvo C, Lawrence D, Hayward M, Yap J, Roberts N, Sheikh A, Kolvekar S, Hausenloy DJ, Yellon DM. Effect of remote ischaemic preconditioning on clinical outcomes in patients undergoing cardiac bypass surgery: a randomised controlled clinical trial. Heart. 2015 Feb;101(3):185-92. doi: 10.1136/heartjnl-2014-306178. Epub 2014 Sep 24. PMID 25252696